CLINICAL TRIAL: NCT00898300
Title: Establishment of a Head and Neck Cancer Tissue/Specimen Bank
Brief Title: Collecting and Storing Tissue Samples From Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: RTOG 0514; CDR0000460036
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; stage I basal cell carcinoma of the lip; stage II basal cell carcinoma of the lip; stage III basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; stage I mucoepidermoid carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage I verrucous carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; stage I adenoid cystic carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; metastatic squamous neck cancer with occult primary; stage I lymphoepithelioma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent adenoid cystic carcinoma of the oral cavity; recurrent basal cell carcinoma of the lip; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent lymphoepithelioma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent salivary gland cancer; recurrent verrucous carcinoma of the larynx; recurrent verrucous carcinoma of the oral cavity; recurrent metastatic squamous neck cancer with occult primary
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Fresh frozen specimens of normal squamous mucosa, tumors, and pre-malignant lesions of the upper aerodigestive tract. 2. Paraffin-embedded tissue sections from head and neck premalignant and malignant lesions. 3. Serum, plasma and isolate lymphocytes from blood drawn from patients with head and neck cancer. 4. Buccal scrapings and saliva samples from patients with head and neck cancer.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with confirmed or suspected head and neck cancer
  Interventions: Other: biologic sample preservation procedure; Procedure: biopsy

INTERVENTIONS:
Other: biologic sample preservation procedure
Procedure: biopsy

SUMMARY:
RATIONALE: Collecting and storing samples of tissue, blood, and saliva from patients with cancer to study in the laboratory may help the study of cancer in the future.

PURPOSE: This laboratory study is collecting and storing tissue samples from patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Establish a tissue/specimen bank of biologic specimens collected from patients with proven or suspected head and neck cancer.
* Establish a database to link materials acquisition and pathologic and clinical information on these patients.
* Correlate clinical-pathological findings on these patients with future scientific studies using the patient database.
* Test new hypotheses as they emerge.

OUTLINE: This is a prospective, multicenter study.

Patients enrolled on active Radiation Therapy Oncology Group clinical trials undergo biopsy or surgical resection of head and neck tumors or premalignant lesions at participating institutions. Tissue and other specimens collected at the time of biopsy or surgery are submitted to the Head and Neck Cancer Tissue/Specimen Bank which acts as a central repository for processing, storing, and preserving patient specimens for translational research. Tissue samples include paraffin-embedded blocks or fresh or frozen samples of normal squamous mucosa, tumors, or premalignant lesions of the upper aerodigestive tract. Other specimens for tissue banking include serum, plasma, and lymphocytes isolated from peripheral blood, as well as samples of patient saliva. Cells obtained from tissue bank specimens may also be used to establish cell lines for future research.

PROJECTED ACCRUAL: An unlimited number of specimens will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed or suspected head and neck cancer

  * Primary site recurrence allowed
* Potentially eligible for or participating in an active Radiation Therapy Oncology Group treatment clinical trial

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent radiotherapy, drug therapy, biopsy, or surgery allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed or suspected head and neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2005-09; Primary Completion 2010-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Establishment of a Head and Neck Cancer Tissue/Specimen Bank | From the start of enrollment to the end of enrollment; enrollment closed at 351 patients

CONTACTS AND LOCATIONS:
Overall Officials: Randal S. Weber, MD, Study Chair — M.D. Anderson Cancer Center
Locations (98):
- United States (97):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - University of California Davis Cancer Center, Sacramento, California
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Winship Cancer Institute of Emory University, Altanta, Georgia
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Good Samaritan Cancer Care Center at Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - St. Vincent Oncology Center, Indianapolis, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Menorah Medical Center, Overland Park, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wood County Oncology Center, Bowling Green, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- McGill Cancer Centre at McGill University, Montreal, Quebec, Canada